CLINICAL TRIAL: NCT05094154
Title: Effect of Antibiotic Choice On ReNal Outcomes (ACORN)
Acronym: ACORN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, EDDIE QIAN, Principal Investigator, Clinical Fellow, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 210591
Record Dates: First submitted 2021-10-22; First posted 2021-10-26 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Sepsis; AKI; Neurotoxicity
MeSH Terms: conditions — Sepsis; Neurotoxicity Syndromes

STUDY DESIGN:
Intervention Model Description: This study will be performed as a pragmatic, randomized controlled clinical trial with parallel group assignment.
Who Masked: Outcomes Assessor
Masking Description: Patients and providers will necessarily be unblinded, but outcomes will be analyzed by a blind assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- anti-pseudomonal cephalosporin (Active Comparator): Participants in the anti-pseudomonal cephalosporin arm will receive at least one dose of an anti-pseudomonal cephalosporin.
  Interventions: Drug: anti-pseudomonal cephalosporin
- anti-pseudomonal penicillin (Active Comparator): Participants in the anti-pseudomonal penicillin arm will receive at least one dose of an anti-pseudomonal penicillin.
  Interventions: Drug: anti-pseudomonal penicillin

INTERVENTIONS:
Drug: anti-pseudomonal cephalosporin — Providers will be prompted to order an anti-pseudomonal cephalosporin, such as cefepime with a dose range of 500 mg, 1,000 mg, or 2,000 mg, and frequency every 6, 8, 12, or 24 hours based on provider discretion.
  Arms: anti-pseudomonal cephalosporin
Drug: anti-pseudomonal penicillin — Providers will be prompted to order anti-pseudomonal penicillin, such as piperacillin-tazobactam with a dose range of 3.375 g or 4.5 g and frequency every 6, 8, or 12 hours based on provider discretion.
  Arms: anti-pseudomonal penicillin

SUMMARY:
Sepsis is one of the most common causes of acute illness and death in the United States. Early, empiric broad-spectrum antibiotics are a mainstay of sepsis treatment. Two classes of antibiotics with activity against Pseudomonas, anti-pseudomonal cephalosporins and anti-pseudomonal penicillins, are commonly used for acutely ill adults with sepsis in current practice. Recent observational studies, however, have raised concern that anti-pseudomonal penicillins may cause renal toxicity. Anti-pseudomonal cephalosporins, by comparison, may be associated with a risk of neurotoxicity. Rigorous, prospective data regarding the comparative effectiveness and toxicity of these two classes of medications among acutely ill patients are lacking. The investigator propose a randomized trial comparing the impact of anti-pseudomonal cephalosporins and anti-pseudomonal penicillins on renal outcomes of acutely ill patients.

DETAILED DESCRIPTION:
Sepsis is a common condition associated with high mortality and morbidity. Antibiotics are an integral component of the management of patients with sepsis. Each hour delay in antibiotic administration in sepsis is associated with an increase in mortality. Clinical guidelines recommend early management bundles, including early broad-spectrum antibiotics, for patients with presumed sepsis in the emergency department and intensive care unit. Since the specific organism causing an infection is rarely known at clinical presentation, empiric broad-spectrum antibiotics are commonly prescribed. For patients at risk for resistant organisms, the most common regimens include vancomycin (to cover gram-positive organisms including methicillin-resistant Staphylococcus aureus) and an anti-pseudomonal cephalosporin or anti-pseudomonal penicillin (to cover gram-negative organisms including Pseudomonas).

Cephalosporins and penicillins are beta-lactam antibiotics that act by inhibiting the synthesis of the peptidoglycan layer of bacterial cell walls. They are commonly used for a variety of infections including empiric broad spectrum coverage for sepsis and suspected nosocomial infections. Several cephalosporins and penicillins have anti-pseudomonal activity, including cefepime, a fourth-generation cephalosporin, ceftazidime, a third-generation cephalosporin, and piperacillin-tazobactam, an extended-spectrum penicillin with beta-lactamase inhibitor. Anti-pseudomonal penicillins are the preferred agents for empiric broad spectrum coverage at many centers, and piperacillin-tazobactam, specifically, has the added benefit of treating anaerobic organisms.

Acute Kidney Injury (AKI) is a common complication of ICU admission. AKI is associated with a six to eight fold increase in mortality in ICU populations is therefore a common target of critical care trials. Sepsis is the most common cause of AKI and accounts for 40-50% of AKI in the intensive care unit (ICU). As the primary treatment for the underlying cause of sepsis, antibiotics are a critical treatment for acutely ill patients, but antibiotics may cause renal injury, and renally-cleared antibiotics may reach supratherapeutic levels in the setting of AKI. Vancomycin has long been associated with AKI. Recently, a number of retrospective observational analyses have examined a potential association between the concurrent administration of vancomycin and piperacillin-tazobactam and the development of AKI, compared with vancomycin alone. These data, however, are likely to be confounded by indication bias and studies evaluating whether piperacillin-tazobactam causes more AKI than other anti-pseudomonal antibiotics have been inconclusive.

Based on this preliminary, observational data, however, some institutions have elected to change their preferred broad spectrum antibiotic regimens from one including an anti-pseudomonal penicillin to one including an anti-pseudomonal cephalosporin. However, others have argued against this approach given the lack of randomized trials comparing the relative efficacy and safety of the two agents as well as observational data suggesting that cephalosporins may be associated with neuro-toxicity.

Tens of thousands of patients each year receive either anti-pseudomonal cephalosporins and penicillins, but no randomized trials have ever compared their relative effectiveness or safety. Each class of medications has been hypothesized to have toxicities that may be relevant for acutely ill patients. Because the relationship between antibiotic choice (anti-pseudomonal cephalosporins or anti-pseudomonal penicillins) and clinically relevant outcomes, such as AKI, are unknown, clinical trial data is urgently needed. Rigorous high-quality evidence that anti-pseudomonal cephalosporins, compared to anti-pseudomonal penicillins, decreases, increases or has no impact on the risk of AKI would have the potential to change the care received by thousands of acutely ill adults each year.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Located in a participating emergency department or medical intensive care unit
* Less than 12 hours from presentation to study hospital
* Treating clinician initiating an order for an anti-pseudomonal cephalosporin or anti-pseudomonal penicillin

Exclusion Criteria:

* Known receipt of > 1 dose of an anti-pseudomonal cephalosporin or anti-pseudomonal penicillin during the last 7 days
* Current documented allergy to cephalosporins or penicillin
* Known to be a prisoner
* Treating clinicians feel that either an anti-pseudomonal cephalosporin or anti-pseudomonal penicillin is required or contraindicated for the optimal treatment of the patient, including for more directed antibiotic therapy against known prior resistant infections or suspected sepsis with an associated central nervous system infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2634 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward T Qian, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported will be made available (including data dictionaries) after de-identification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available 3 months following publication of outcomes and will remain available for at least 5 years.
Access Criteria: Data will be made available to researchers who provide a methodologically sound proposal that has been approved by the Vanderbilt Institutional Review Board and the study executive committee.

REFERENCES:
- [Background] Cecconi M, Evans L, Levy M, Rhodes A. Sepsis and septic shock. Lancet. 2018 Jul 7;392(10141):75-87. doi: 10.1016/S0140-6736(18)30696-2. Epub 2018 Jun 21. PMID 29937192
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Liu VX, Fielding-Singh V, Greene JD, Baker JM, Iwashyna TJ, Bhattacharya J, Escobar GJ. The Timing of Early Antibiotics and Hospital Mortality in Sepsis. Am J Respir Crit Care Med. 2017 Oct 1;196(7):856-863. doi: 10.1164/rccm.201609-1848OC. PMID 28345952
- [Background] Damiani E, Donati A, Serafini G, Rinaldi L, Adrario E, Pelaia P, Busani S, Girardis M. Effect of performance improvement programs on compliance with sepsis bundles and mortality: a systematic review and meta-analysis of observational studies. PLoS One. 2015 May 6;10(5):e0125827. doi: 10.1371/journal.pone.0125827. eCollection 2015. PMID 25946168
- [Background] Thakar CV, Christianson A, Freyberg R, Almenoff P, Render ML. Incidence and outcomes of acute kidney injury in intensive care units: a Veterans Administration study. Crit Care Med. 2009 Sep;37(9):2552-8. doi: 10.1097/CCM.0b013e3181a5906f. PMID 19602973
- [Background] Uchino S, Kellum JA, Bellomo R, Doig GS, Morimatsu H, Morgera S, Schetz M, Tan I, Bouman C, Macedo E, Gibney N, Tolwani A, Ronco C; Beginning and Ending Supportive Therapy for the Kidney (BEST Kidney) Investigators. Acute renal failure in critically ill patients: a multinational, multicenter study. JAMA. 2005 Aug 17;294(7):813-8. doi: 10.1001/jama.294.7.813. PMID 16106006
- [Background] Hoste EA, Bagshaw SM, Bellomo R, Cely CM, Colman R, Cruz DN, Edipidis K, Forni LG, Gomersall CD, Govil D, Honore PM, Joannes-Boyau O, Joannidis M, Korhonen AM, Lavrentieva A, Mehta RL, Palevsky P, Roessler E, Ronco C, Uchino S, Vazquez JA, Vidal Andrade E, Webb S, Kellum JA. Epidemiology of acute kidney injury in critically ill patients: the multinational AKI-EPI study. Intensive Care Med. 2015 Aug;41(8):1411-23. doi: 10.1007/s00134-015-3934-7. Epub 2015 Jul 11. PMID 26162677
- [Background] Gomez H, Kellum JA. Sepsis-induced acute kidney injury. Curr Opin Crit Care. 2016 Dec;22(6):546-553. doi: 10.1097/MCC.0000000000000356. PMID 27661757
- [Background] Arnaud FCS, Liborio AB. Attributable nephrotoxicity of vancomycin in critically ill patients: a marginal structural model study. J Antimicrob Chemother. 2020 Apr 1;75(4):1031-1037. doi: 10.1093/jac/dkz520. PMID 31904834
- [Background] Filippone EJ, Kraft WK, Farber JL. The Nephrotoxicity of Vancomycin. Clin Pharmacol Ther. 2017 Sep;102(3):459-469. doi: 10.1002/cpt.726. Epub 2017 Jun 5. PMID 28474732
- [Background] Bellos I, Karageorgiou V, Pergialiotis V, Perrea DN. Acute kidney injury following the concurrent administration of antipseudomonal beta-lactams and vancomycin: a network meta-analysis. Clin Microbiol Infect. 2020 Jun;26(6):696-705. doi: 10.1016/j.cmi.2020.03.019. Epub 2020 Mar 25. PMID 32222460
- [Background] Rutter WC, Burgess DR, Talbert JC, Burgess DS. Acute kidney injury in patients treated with vancomycin and piperacillin-tazobactam: A retrospective cohort analysis. J Hosp Med. 2017 Feb;12(2):77-82. doi: 10.12788/jhm.2684. PMID 28182801
- [Background] Carreno J, Smiraglia T, Hunter C, Tobin E, Lomaestro B. Comparative incidence and excess risk of acute kidney injury in hospitalised patients receiving vancomycin and piperacillin/tazobactam in combination or as monotherapy. Int J Antimicrob Agents. 2018 Nov;52(5):643-650. doi: 10.1016/j.ijantimicag.2018.08.001. Epub 2018 Aug 10. PMID 30103003
- [Background] Downes KJ, Cowden C, Laskin BL, Huang YS, Gong W, Bryan M, Fisher BT, Goldstein SL, Zaoutis TE. Association of Acute Kidney Injury With Concomitant Vancomycin and Piperacillin/Tazobactam Treatment Among Hospitalized Children. JAMA Pediatr. 2017 Dec 4;171(12):e173219. doi: 10.1001/jamapediatrics.2017.3219. Epub 2017 Dec 4. PMID 28973124
- [Background] Kalligeros M, Karageorgos SA, Shehadeh F, Zacharioudakis IM, Mylonakis E. The association of acute kidney injury with the concomitant use of vancomycin and piperacillin/tazobactam in children: A systematic review and meta-analysis. Antimicrob Agents Chemother. 2019 Sep 9;63(12):e01572-19. doi: 10.1128/AAC.01572-19. Epub 2019 Oct 7. PMID 31591125
- [Background] O'Callaghan K, Hay K, Lavana J, McNamara JF. Acute kidney injury with combination vancomycin and piperacillin-tazobactam therapy in the ICU: A retrospective cohort study. Int J Antimicrob Agents. 2020 Jul;56(1):106010. doi: 10.1016/j.ijantimicag.2020.106010. Epub 2020 May 12. PMID 32413387
- [Background] Hammond DA, Smith MN, Painter JT, Meena NK, Lusardi K. Comparative Incidence of Acute Kidney Injury in Critically Ill Patients Receiving Vancomycin with Concomitant Piperacillin-Tazobactam or Cefepime: A Retrospective Cohort Study. Pharmacotherapy. 2016 May;36(5):463-71. doi: 10.1002/phar.1738. Epub 2016 Apr 1. PMID 26952639
- [Background] Kang S, Park J, Yu YM, Park MS, Han E, Chang MJ. Comparison of acute kidney injury and clinical prognosis of vancomycin monotherapy and combination therapy with beta-lactams in the intensive care unit. PLoS One. 2019 Jun 5;14(6):e0217908. doi: 10.1371/journal.pone.0217908. eCollection 2019. PMID 31166993
- [Background] Buckley MS, Hartsock NC, Berry AJ, Bikin DS, Richards EC, Yerondopoulos MJ, Kobic E, Wicks LM, Hammond DA. Comparison of acute kidney injury risk associated with vancomycin and concomitant piperacillin/tazobactam or cefepime in the intensive care unit. J Crit Care. 2018 Dec;48:32-38. doi: 10.1016/j.jcrc.2018.08.007. Epub 2018 Aug 11. PMID 30172962
- [Background] Hammond DA, Smith MN, Li C, Hayes SM, Lusardi K, Bookstaver PB. Systematic Review and Meta-Analysis of Acute Kidney Injury Associated with Concomitant Vancomycin and Piperacillin/tazobactam. Clin Infect Dis. 2017 Mar 1;64(5):666-674. doi: 10.1093/cid/ciw811. Epub 2016 Dec 10. PMID 27940946
- [Background] Molina KC, Barletta JF, Hall ST, Yazdani C, Huang V. The Risk of Acute Kidney Injury in Critically Ill Patients Receiving Concomitant Vancomycin With Piperacillin-Tazobactam or Cefepime. J Intensive Care Med. 2020 Dec;35(12):1434-1438. doi: 10.1177/0885066619828290. Epub 2019 Feb 10. PMID 30741072
- [Background] Luther MK, Timbrook TT, Caffrey AR, Dosa D, Lodise TP, LaPlante KL. Vancomycin Plus Piperacillin-Tazobactam and Acute Kidney Injury in Adults: A Systematic Review and Meta-Analysis. Crit Care Med. 2018 Jan;46(1):12-20. doi: 10.1097/CCM.0000000000002769. PMID 29088001
- [Background] Abanades S, Nolla J, Rodriguez-Campello A, Pedro C, Valls A, Farre M. Reversible coma secondary to cefepime neurotoxicity. Ann Pharmacother. 2004 Apr;38(4):606-8. doi: 10.1345/aph.1D322. Epub 2004 Feb 24. PMID 14982986
- [Background] Balderia PG, Chandorkar A, Kim Y, Patnaik S, Sloan J, Newman GC. Dosing Cefepime for Renal Function Does Not Completely Prevent Neurotoxicity in a Patient With Kidney Transplant. J Patient Saf. 2018 Jun;14(2):e33-e34. doi: 10.1097/PTS.0000000000000225. PMID 26102002
- [Derived] Qian ET, Casey JD, Wright A, Wang L, Shotwell MS, Siemann JK, Dear ML, Stollings JL, Lloyd BD, Marvi TK, Seitz KP, Nelson GE, Wright PW, Siew ED, Dennis BM, Wrenn JO, Andereck JW, Han JH, Self WH, Semler MW, Rice TW; Vanderbilt Center for Learning Healthcare and the Pragmatic Critical Care Research Group. Cefepime vs Piperacillin-Tazobactam in Adults Hospitalized With Acute Infection: The ACORN Randomized Clinical Trial. JAMA. 2023 Oct 24;330(16):1557-1567. doi: 10.1001/jama.2023.20583. PMID 37837651
- [Derived] Qian ET, Casey JD, Wright A, Wang L, Siemann J, Dear ML, Stollings J, Lloyd BD, Seitz K, Nelson G, Wright P, Siew ED, Dennis B, Wrenn J, Andereck J, Self WH, Semler MW, Rice TW; Vanderbilt Learning Healthcare System Platform Investigators. Protocol and statistical analysis plan for the Antibiotic Choice On ReNal outcomes (ACORN) randomised clinical trial. BMJ Open. 2023 Mar 10;13(3):e066995. doi: 10.1136/bmjopen-2022-066995. PMID 36898748

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Among 3,806 patients who met inclusion criteria, 1,172 were excluded. Of the 2,634 enrolled and randomized, 4 were prisoners and excluded post-randomization from subsequent data collection and analysis, 119 did not receive a dose of anti-pseudomonal cephalosporin or anti-pseudomonal penicillin in the 7 days after enrollment and were not included in the primary analysis, leaving 2,511 included in the primary analysis. Thus 2,511 matches the number reported in the Study Design section.
Period: Overall Study
Arm/Group | Anti-pseudomonal Cephalosporin | Anti-pseudomonal Penicillin
Started | 1277 | 1357
Completed | 1214 | 1297
Not Completed | 63 | 60
Not completed — Participants experiencing incarceration or involuntary detainment. | 3 | 1
Not completed — Did not receive appropriate drug in 7 days post-enrollment. | 60 | 59

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti-pseudomonal Cephalosporin | Anti-pseudomonal Penicillin | Total
Number analyzed (Participants) | 1214 | 1297 | 2511
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: One value was missing for a participant in the anti-pseudomonal penicillin group.
  years
    number analyzed (Participants) | 1214 | 1296 | 2510
    (all) | 57 [42 to 68] | 59 [44 to 69] | 58 [43 to 69]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One value was missing for a participant in the anti-pseudomonal penicillin group.
  Participants
    number analyzed (Participants) | 1214 | 1296 | 2510
    Female | 523 | 548 | 1071
    Male | 691 | 748 | 1439
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 28 values were unknown for participants in the anti-pseudomonal cephalosporin group and 33 values were unknown for participants in anti-pseudomonal penicillin group.
  Participants
    Race and Ethnicity: number analyzed (Participants) | 1186 | 1264 | 2450
    Race and Ethnicity: White, non-Hispanic | 913 | 950 | 1863
    Race and Ethnicity: Black, non-Hispanic | 190 | 209 | 399
    Race and Ethnicity: Hispanic | 59 | 73 | 132
    Race and Ethnicity: Other | 24 | 32 | 56
Region of Enrollment [Number; unit: participants]
  United States | 1214 | 1297 | 2511

OUTCOME MEASURES:

1. Primary Outcome: Acute Kidney Injury (AKI) Ordinal Scale
Description: Acute Kidney Injury Score between randomization and day 14. The acute kidney injury score is an ordinal outcome containing the stages of AKI as defined by Kidney Disease: Improving Global Outcomes (KDIGO) creatinine criteria, new renal replacement therapy (RRT), and death:
  0 = No AKI
  1. = Stage 1 AKI (Creatinine increase by 1.5-1.9 times baseline OR increase by >= 0.3 mg/dL)
  2. = Stage 2 AKI (Creatinine increase by 2.0-2.9 times baseline)
  3. = Stage 3 AKI (Creatinine increase by >= 3.0 times baseline OR increase to >= 4.0 mg/dL OR New RRT)
  4. = Death
Time Frame: 14 days post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-pseudomonal Cephalosporin | Anti-pseudomonal Penicillin
Number analyzed (Participants) | 1214 | 1297
Participants
  0 = Survived without AKI | 910 | 952
  1 = Survived with Stage 1 AKI | 86 | 100
  2 = Survived with Stage 2 AKI | 41 | 70
  3 = Survived with Stage 3 AKI | 85 | 97
  4 = Died | 92 | 78

2. Secondary Outcome: Major Adverse Kidney Events Within 14 Days (MAKE14)
Description: Composite outcome of death within 14 days, new renal replacement therapy within 14 days, or stage 2 or higher AKI at day 14
Time Frame: 14 days post-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Anti-pseudomonal Cephalosporin | Anti-pseudomonal Penicillin
Number analyzed (Participants) | 1214 | 1297
Participants | 124 | 114

3. Secondary Outcome: Delirium and Coma-Free Days to Day 14
Description: The number of days alive and free of coma and delirium in the 14 days after enrollment
Time Frame: 14 days post-enrollment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Anti-pseudomonal Cephalosporin | Anti-pseudomonal Penicillin
Number analyzed (Participants) | 1214 | 1297
days | 14 [14 to 14] | 14 [14 to 14]

4. Other Pre Specified Outcome: Post-Emergency Department Disposition
Description: Patient disposition (ex. floor unit or intensive care unit) at day 14 post-enrollment from the emergency department.
Time Frame: 14 days post-enrollment
Measure: Number; unit: participants
Arm/Group | Anti-pseudomonal Cephalosporin | Anti-pseudomonal Penicillin
Number analyzed (Participants) | 1135 | 1243
participants
  Home | 26 | 23
  Ward | 1016 | 1117
  ICU | 93 | 103

ADVERSE EVENTS:
Time Frame: 28 days.
Description: Per the protocol and SAP, the primary, secondary, and exploratory outcomes were reported as clinical outcomes not as AEs unless the event was Definitely Related or Probably or Possibly Related to the study.
  ONLY the following types of AEs were collected, recorded, and reportable:
  * AEs that are Serious and Definitely Related, Probably or Possibly Related, or of Uncertain Relationship.
  * AEs that are Unexpected and Definitely Related, Probably or Possibly Related, or of Uncertain Relationship.
Arm/Group | Anti-pseudomonal Cephalosporin | Anti-pseudomonal Penicillin
All-Cause Mortality (participants affected / at risk) | 104/1214 | 106/1297
Serious Adverse Events (participants affected / at risk) | 0/1214 | 0/1297
Other Adverse Events (participants affected / at risk) | 0/1214 | 1/1297
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anti-pseudomonal Cephalosporin (N=1214) | Anti-pseudomonal Penicillin (N=1297)
Blood product related allergy (Immune system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT05094154/Prot_SAP_000.pdf